CLINICAL TRIAL: NCT06575101
Title: Resting Energy Expenditure and Substrate Consumption in Cardiac Arrest Patients Under Target Temperature Management
Status: Recruiting | Type: Observational
Sponsor: Tang Ziren (Other)
Responsible Party: Sponsor-Investigator, Tang Ziren, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Other Study IDs: 2024-4-15-1
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Targeted Temperature Management; Cardiac Arrest; Resting Energy Expenditure; Nutrition
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 33℃ group
  Interventions: Procedure: Target Temperature Management Treatment
- 36℃ group
  Interventions: Procedure: Target Temperature Management Treatment

INTERVENTIONS:
Procedure: Target Temperature Management Treatment — Target Temperature Management Treatment

SUMMARY:
This study is a single-center, prospective, observational study. According to the sample size formula, an estimated 40 cases should be collected, all of whom are from the emergency intensive care unit. After successful cardiopulmonary resuscitation, the enrolled patients will be transferred to the emergency intensive care unit for further standardized target temperature management (TTM). They will be divided into 33 ° C hypothermia group and 36 ° C hypothermia group according to the patient's core body temperature. The baseline data of the patients will be collected at the beginning. After admission to the hospital, they were fasted within 24 hours to reach the target temperature, and then 20kcal/kg/d parenteral nutrition will be given. At selected time points (T0: the initial time point before TTM; T1: the core temperature was reduced to 33 ° C or 36 ° C; T2-T4: 33 ° C or 36 ° C was maintained for 24h, 48h, 72h; T5: the end of rewarming; Tend: the last REE measurement before discharge or death) , various observation indicators will be collected, including resting energy expenditure (REE), glucose oxidation rate, fat oxidation rate, protein oxidation rate, and metabolism of three major nutrients Proportion. Neurological outcomes were followed up 28 days after onset according to the Cerebral Performance Categories (CPC) score.

ELIGIBILITY:
Inclusion Criteria:

* Be admitted to the emergency department of Beijing Chao-yang Hospital, Capital Medical University;
* Successfully resuscitated, and are unconscious after restoration of spontaneous circulation (ROSC);
* Be admitted to the intensive care unit (ICU) for advanced life support such as endotracheal intubation after restoration of spontaneous circulation (ROSC);
* Accepted target temperature management (TTM) therapy after restoration of spontaneous circulation (ROSC);

Exclusion Criteria:

* Age > 18 years old；
* Incomplete clinical data and loss of follow-up;
* Traumatic brain injury or cerebrovascular accident revealed by computed tomography (CT)；
* Severe metabolic abnormalities are known: cachexia, thyroid dysfunction, and cancer；
* Indirect calorimetry measurement is not possible such as sustained oxygen concentration > 70%；
* There were no signs of resuscitation at the time of admission；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients(age >18 years) who have been successfully resuscitated from cardiac arrest who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Resting Energy Expenditure | 7 days
  The primary outcome measure is the changes resting energy expenditure(REE) in the patients at various time points.
  patients at various time points.
Glucose oxidation rate | 7 days
  The primary outcome measure is the statistical differences in Glucose oxidation rate between the two groups of patients at various time points.
Fat oxidation rate | 7 days
  The primary outcome measure is the statistical differences in fat oxidation rate between the two groups of patients at various time points.
Protein oxidation rate | 7 days
  The primary outcome measure is the statistical differences in protein oxidation rate between the two groups of patients at various time points.
Metabolic supply proportion of glucose, fat, protein | 7 days
  The primary outcome measure is the statistical differences in metabolic supply proportion of glucose, fat, protein (measuring by indirect calorimetry) between the two groups of patients at various time points.

SECONDARY OUTCOMES:
CPC score | 28 days
  CPC = Cerebral Performance Category Score.There are 5 levels of CPC score. CPC 1-2 means good prognosis of neurological function, CPC3-5 means bad prognosis of neurological function. The Secondary Outcome of the study is the statistical differences in the proportion of patients with good neurological outcome(CPC1-2) in the two groups at 28 days after CA.
Mortality rate | 28 days
  The Secondary Outcome of the study is the statistical differences in the mortality rate of two groups at 28 days after CA.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing chao-yang Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: The identified survey data will be made available for research purposes by contacting the corresponding authors